CLINICAL TRIAL: NCT04310605
Title: Cognitive Behaviour Therapy (CBT) for Tinnitus Treatment: Implementation and Validity
Brief Title: Effectiveness of Specialised Cognitive Behavioural Therapy (CBT) for Tinnitus.
Status: Completed | Type: Observational
Sponsor: Maastricht University (Other)
Collaborators: SWOL Limburgs Fonds voor Revalidatie (Unknown); Flemish Government, Belgium (Unknown); The Netherlands Organization for Scientific Research (NWO) (Unknown); Libra Revalidatie en Audiologie (Unknown)
Responsible Party: Sponsor
Other Study IDs: ECP-152 05_12_2014
Record Dates: First submitted 2020-03-13; First posted 2020-03-17 (Actual); Last update posted 2020-03-17 (Actual); Status verified 2020-03

CONDITIONS: Tinnitus, Subjective
Keywords: tinnitus; CBT; cognitive behaviour therapy
MeSH Terms: conditions — Tinnitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Step 1 only: Participants in the study who only receive Step 1 of specialised CBT
  Interventions: Behavioral: CBT 1
- Step 1 and 2: Participants who receive both Step 1 and Step 2 of speciliased CBT for tinnitus.
  Interventions: Behavioral: CBT 1; Behavioral: CBT 2

INTERVENTIONS:
Behavioral: CBT 1 — CBT for tinnitus (Step 1) comprised: individual audiometric assessment, and counselling about hearing and tinnitus (1hr) with an audiologist; a one-off educational group session (a max 10 participants and partners) (2hrs); an assessment session with a psychologists (1 hr).
Behavioral: CBT 2 — Step 2 group sessions were 2 hrs long over a 12-week period. Two therapists (a psychologist and physiotherapist) were present at any one time for Step 2 sessions. Step 2 included: psycho-education; exposure therapy; mindfulness exercises; cognitive restructuring; attention redirecting techniques; stress reduction; and, relaxation techniques. Evening sessions were also provided for participants to attend with family or partners.
  Groups: Step 1 and 2

SUMMARY:
This is an observational study of specialised CBT for tinnitus for adults delivered in routine care.

ELIGIBILITY:
Inclusion Criteria:

* Tinnitus is the primary complaint and reason for seeking help
* Participant is at least 17 years of age,

Exclusion Criteria:

* Unable to read and write in Dutch
* Tinnitus is not the primary complaint
* Person is under 17 years of age
* Participant has a health condition that prevents them from attending treatment centre
* An Ear Nose Throat (ENT) physician assesses the participant as having ontological condition that requires medical treatment

Min Age: 17 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Adults with tinnitus
Sampling Method: Non-Probability Sample
Enrollment: 403 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2016-11-16 (Actual); Study Completion 2016-11-16 (Actual)

PRIMARY OUTCOMES:
Health Utilities Index-III | 12 months
  The Health Utilities Index (HUI; Feeny et al., 2002; Horsman, Furlong, Feeny, & Torrance, 2003) is a 17-item measure designed to assess health related quality of life.

SECONDARY OUTCOMES:
Tinnitus Handicap Inventory (THI) | 12 months
  The THI (Newman, Jacobson, & Spitzer, 1996; Newman, Sandridge, & Jacobson, 1998).is a 25 items measure of the impact of tinnitus on daily life that includes three subscales. The subscales cover functional (mental, social/occupational and physical functioning), emotional impact and catastrophic responses to tinnitus.
Hospital Anxiety and Depression Scale (HADS; Zigmond & Snaith, 1983). | 12 months
  The HADS is a widely used measure of psychological distress in people experiencing a concurrent physical health condition. It has 14 items and respondents use a Likert-type scale to indicate how often they have had a particular feeling in the previous week (e.g. "I feel tense or wound up").
Tinnitus Catastrophizing Scale (TCS) | 12 months
  Tinnitus Catastrophizing Scale (TCS; Cima, Crombez, & Vlaeyen, 2011). The TCS was used to assess the degree to which people thought or expected the worst about tinnitus (i.e. catastrophizing). The TCS is a 13-item measure based on the Pain Catastrophizing Scale (Sullivan, Bishop, & Pivik, 1995) and respondents use a five point scale to indicate the degree to which statements applies to them (e.g. It's terrible and I think it's never going to get any better). The total score on the TCS ranges from 0 to 65.
Fear of Tinnitus Questionnaire (FTQ) | 12 months
  The FTQ is a 17-item self-report measure intended and designed to assess respondents' level of fear regarding their tinnitus. Items in the questionnaire are presented as a series of statements (e.g. "I am afraid that my tinnitus will become worse") from which respondents are asked to indicate if it is applicable to their current situation. Each statement receives a score of 1 when applicable. The total score is the sum of all applicable statements and provides an overall rating of fear of tinnitus and ranges from 0 to 17.
Tinnitus Questionnaire (TQ) | 12 months
  The Tinnitus Questionnaire (TQ; Hallam, Jakes, & Hinchcliffe, 1988) is a self-report questionnaire designed to asses distress and interference in daily activities that is associated with tinnitus. It has 52 items and uses a three-point scale to indicate levels of distress on six subscales. The total possible score on the TQ ranges from 0-84.
Tinnitus Disability Index (TDI) | 12 months
  The Tinnitus Disability Index (TDI; Cima, Vlaeyen, Maes, Joore, & Anteunis, 2011) is a seven-item self-report questionnaire that assesses the level of interferences in daily activities (such as occupational, social, and recreational) attributed to tinnitus. Respondents use an 11-point scale to indicate the level of interference ranging from 0 no disability, to 10 total disability. The total score ranges from 0 to 70 with higher scores indicating higher levels of interference.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Cima RF, Maes IH, Joore MA, Scheyen DJ, El Refaie A, Baguley DM, Anteunis LJ, van Breukelen GJ, Vlaeyen JW. Specialised treatment based on cognitive behaviour therapy versus usual care for tinnitus: a randomised controlled trial. Lancet. 2012 May 26;379(9830):1951-9. doi: 10.1016/S0140-6736(12)60469-3. PMID 22633033